CLINICAL TRIAL: NCT01817803
Title: A Prospective, Single-center, Open-label, Pilot Study to Compare the Effectiveness and Safety of Diuretics Add-On Strategy in Chronic Heart Failure Patients (DIOS 1)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0013
Record Dates: First submitted 2013-03-20; First posted 2013-03-25 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Congestive Heart Failure
Keywords: Heart failure; diuretics; kidney; glomerular filtration rate
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Spironolactone; Metolazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1) Add furosemide/no spironolactone (Active Comparator)
  Interventions: Drug: furosemide/no spironolactone
- 2) Add metolazone/no spironolactone (Active Comparator)
  Interventions: Drug: metolazone/no spironolactone
- 3) Add furosemide/spironolactone (Active Comparator)
  Interventions: Drug: furosemid/spironolactone
- 4) Add metolazone/spironolactone (Active Comparator)
  Interventions: Drug: metolazone/spironolactone

INTERVENTIONS:
Drug: furosemide/no spironolactone — furosemide (doubling previous furosemide dose)
  Arms: 1) Add furosemide/no spironolactone
Drug: metolazone/no spironolactone — metolazone (add 2.5mg qod)
  Arms: 2) Add metolazone/no spironolactone
Drug: furosemid/spironolactone — furosemide (doubling previous furosemide dose)+spironolactone (doubling previous spironolactone dose or add 12.5mg BID if previous non-user)
  Arms: 3) Add furosemide/spironolactone
Drug: metolazone/spironolactone — metolazone (add 2.5mg qod)+ spironolactone (doubling previous spironolactone dose or add 12.5mg BID if previous non-user)
  Arms: 4) Add metolazone/spironolactone

SUMMARY:
To compare the effectiveness and safety of diuretics add-on strategy in chronic heart failure patients

ELIGIBILITY:
Inclusion Criteria:

1. dyspnea at rest or minimal activity
2. tachypnea (respiratory rate > 20/min) or rales or pulmonary edema on chest X-ray
3. who need diuretics add over 40mg of daily furosemide dose

Exclusion Criteria:

1. Hospitalization for acute heart failure decompensation
2. cardiogenic shock (Systolic Blood Pressure < 80mmHg)
3. Need or plan for renal replacement therapy (dialysis, kidney transplant)
4. serum creatine level > 2.5mg/dl
5. serum potassium (K+) > 5.5mg/dl
6. daily spironolactone dose > 50mg
7. previous thiazide or metolazone user
8. Age > 75 years old or poor compliance patients 9. allergy, adverse drug reaction, hypersensitivity to any kinds of diuretics 10. life expectancy < 6 months (e.g. metastatic malignancy, liver cirrhosis) 11. pregnancy or women at age of childbearing potential

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
efficacy and safety of diuretics add-on strategy | D+0, D+7, D+30, D+90
  1) body weight change, symptoms & signs change, systemic impedance change 2) serum & urine creatinine change, serum & urine electrolyte change, biomarkers change, clinical outcomes ( all-cause mortality, all-cause rehospitalization, start of renal replacement therapy)